CLINICAL TRIAL: NCT04122521
Title: Prospective Observational Study of Imaging-based Prediction for Genomic Mutations and Prognosis in Glioma
Brief Title: Radiogenomic and Prognosis Analysis in Glioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Sung Kim, Professor, Asan Medical Center
Other Study IDs: AsanMCHSKim_03
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pathologic specimen with next generation sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glioma: Patients suspected of glioma
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI

SUMMARY:
This study aims to evaluate whether MRI can be used to predict genomics and prognosis in glioma. Given the profound prognostic significance of genetic mutations seen in glioma, there have been increasing attempts to correlate imaging characteristics with genetic, mutational and expression patterns. To be able to predict genomics and prognosis based on imaging alone will prove useful in patients with involvement of glioma in delicate areas of the brain and better reflect tumor and molecular heterogeneity.

DETAILED DESCRIPTION:
Previous studies have proposed certain imaging characteristics correlating with genetic, molecular and expression patterns. Advanced imaging provides additional clues but no studies have examined its added value particularly in a prospective setting. The investigator's aim to evaluate preoperative MRI for patients suspected of glioma to predict IDH mutation, 1p19q codeletion, MGMT methylation and EGFR mutation status using imaging characteristics such as margin, patterns of contrast enhancement and edema as well as diffusion and perfusion characteristics. This will be confirmed pathologically and further correlated with patients' long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of glioma undergoing MRI examination prior to surgery
* MRI including advanced imaging such as cerebral blood volume, apparent diffusion coefficient and amide proton transfer imaging
* Signed informed consent

Exclusion Criteria:

* Pathologic confirmation as tumors other than glioma
* Patients who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulates, electronic infusion pumps, etc), because such devices may be displaced or malfunction
* Patients who are pregnant or breast feeding; urine pregnancy test will be performed on women of child bearing potential

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of tertiary hospital center
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2020-01-12 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Time to progression | Through study completion, an average of 2 years
  The response was determined by a modification of the response assessment in neuro-oncology (RANO) criteria that combined the image assessment, neurologic evaluation and assessment of steroid use.

SECONDARY OUTCOMES:
Genomics including IDH mutation, 1p19q codeletion, MGMT methylation and EGFR mutation status | 2 months
  Proportion of positive IDH mutation, 1p19q codeletion, MGMT methylation and EGFR mutation in percentage (%)
Progression free survival | Through study completion, an average of 3 years
  Estimated probable duration of life without disease progression, from on-study date to earlier progression date or date of death from any cause, using the Kaplan-Meier method with censoring. The response was determined by a modification of the RANO criteria that combined the image assessment, neurologic evaluation and assessment of steroid use.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sung Kim, MD PhD, Principal Investigator — Asan Medical Center; Ji Eun Park, MD PhD, Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes